CLINICAL TRIAL: NCT04261296
Title: Comparison of the Efficacy of Dry Needling and Balneotherapy in the Treatment of Myofascial Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ahi Evran University Education and Research Hospital (Other)
Responsible Party: Principal Investigator, Zeynep Karakuzu Güngör, Research Assistant, Ahi Evran University Education and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019-22/217
Record Dates: First submitted 2020-02-04; First posted 2020-02-07 (Actual); Last update posted 2023-03-01 (Actual); Status verified 2023-02

CONDITIONS: Myofascial Pain Syndrome of Neck
Keywords: dry needling; spa
MeSH Terms: interventions — Dry Needling; Balneology

STUDY DESIGN:
Intervention Model Description: randomized controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dry needling (Experimental): Arm 1: Dry needling group. Dry needling will be done with painful trigger point and it will be waited for about 20 minutes. This treatment will be repeated once a week for 3 weeks.No medication is used in this treatment.
  Interventions: Other: dry needling
- balneotherapy (Experimental): Arm 2: Balneotherapy A total of 15 sessions, 20 minutes a day, 5 days a week for 3 weeks, will be held in the spa, which operates within the body of Kırşehir Ahi Evran University Physical Therapy and Rehabilitation Center.
  Interventions: Other: balneotherapy
- Dry needling + balneotherapy (Experimental): Arm3: dry needling + balneotherapy Both of these methods will be applied to patients in the third group.
  Interventions: Other: dry needling +balneotherapy

INTERVENTIONS:
Other: dry needling — In this treatment, depending on the thickness of the adipose tissue under the skin, 13 mm, 25 mm or 30 mm long; 0.20 mm thick acupuncture needle is used
  Arms: Dry needling
Other: balneotherapy — This treatment method; An "alert-fit" performed in a certain time interval and in a cure style by using the methods and doses of hot mineral waters, gases and peloids (sludge) from natural underground, determined in detail, repeatedly in series as bath, drinking and inhalation treatments. treatment can be defined as. There are studies showing that the effect of balneotherapy is mechanical, thermal, chemical, anti-inflammatory and immunological.
  Other Names: Spa
  Arms: balneotherapy
Other: dry needling +balneotherapy — Both of these methods will be applied to patients in the third group.
  Arms: Dry needling + balneotherapy

SUMMARY:
Myofascial pain syndrome (MAS) is a syndrome characterized by muscle spasm, tenderness, limited range of motion, stiffness, fatigue and sometimes autonomic dysfunctions accompanying pain and pain caused by trigger points in the tense bands formed in the muscles The disease is diagnosed clinically and there are many pharmacological and non-pharmacological approaches in treatment.

One of these treatments is dry needle therapy. Dry needling has been used for a long time in the treatment of myofascial pain syndrome.

Another treatment used in the treatment of myofascial pain syndrome is balneotherapy (spa treatment At Ahi Evran University Physical Therapy and Rehabilitation Center, balneotherapy is frequently used in the treatment of patients with myofascial pain syndrome.

The aim of this study is to compare the effectiveness of dry needling and balneotherapy, which has been used in the treatment of myofascial pain syndrome for many years.

DETAILED DESCRIPTION:
Myofascial pain syndrome (MAS) is a syndrome characterized by muscle spasm, tenderness, limited range of motion, stiffness, fatigue and sometimes autonomic dysfunctions accompanying pain and pain caused by trigger points in the tense bands formed in the muscles The disease is diagnosed clinically and there are many pharmacological and non-pharmacological approaches in treatment.

One of these treatments is dry needle therapy. Dry needling has been used for a long time in the treatment of myofascial pain syndrome.

Another treatment used in the treatment of myofascial pain syndrome is balneotherapy (spa treatment At Ahi Evran University Physical Therapy and Rehabilitation Center, balneotherapy is frequently used in the treatment of patients with myofascial pain syndrome.

The aim of this study is to compare the effectiveness of dry needling and balneotherapy, which has been used in the treatment of myofascial pain syndrome for many years.

120 volunteers are planned to be included in this study. Patients will be randomly divided into 3 groups. (randomization will be done as 1: 1: 1 with a closed envelope). The patients in the first group will be given "dry needle treatment" for the aching muscle. No medication is used in this treatment.In this treatment, depending on the thickness of the adipose tissue under the skin, 13 mm, 25 mm or 30 mm long; 0.20 mm thick acupuncture needle is used. Dry needling will be done with painful trigger point and it will be waited for about 20 minutes. This treatment will be repeated once a week for 3 weeks.

Patients in the second group will be given "spa treatment". A total of 15 sessions, 20 minutes a day, 5 days a week for 3 weeks, will be held in the spa, which operates within the body of Kırşehir Ahi Evran University Physical Therapy and Rehabilitation Center. Both of these methods will be applied to patients in the third group.

Evaluations will be repeated before treatment, 1st week after treatment and Week 12 (3rd Month). Patients' neck range of motion (by measuring with goniometer) will be evaluated and pressure pain threshold will be measured using algometer.

Patients' pain levels will be evaluated with Visual Analogue Scale, their moods with Beck Depression Scale, anxiety levels with Beck Anxiety Scale, fear of movement with Tampa Kinesiophobia Scale, neck functions with Neck Disability Questionnaire Questionnaire, and quality of life level with SF-36 Quality of Life Scale.

In addition, the Global Assessment Scale will be used to evaluate patients at the 1st and 12th weeks after treatment. This scale is scored as "-1 = deterioration, 0 = no change, 1 = slight improvement, 2 = significant improvement and 3 = near-normal improvement". Survey applications will take approximately 10 minutes.

ELIGIBILITY:
Inclusion Criteria:

1. Female and male patients between the ages of 18-50 who have been diagnosed as "myofascial pain syndrome (MAS)" by clinical and examination
2. Patients with cooperations who can correctly understand what is stated in the patient information form
3. Patients who consent to participate in the study according to the informed voluntary consent form will be included in the study.

Exclusion Criteria:

1. Presence of cervical disc hernia, radiculopathy or myelopathy
2. Having tumoral, infectious, psychiatric, systemic disease and bleeding diathesis
3. Stage 3-4 osteodegeneration
4. Having a diagnosis of fibromyalgia syndrome according to the diagnostic criteria of 2016 American College of Rheumatology
5. Presence of kyphoscoliosis
6. Pregnancy
7. Having had previous brain, neck or shoulder surgery
8. Having received treatment for MAS in the last 6 months
9. Symptom onset duration is less than 3 months
10. Having analgesic use for any reason
11. Failure to cooperate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2020-02-10 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-05-31 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | Measurements will be made before treatment, at the 1st week after treatment and at the 3rd month after treatment. Then change of the level of pain will be investigated.
  Pain level of the patients will be determined by "Visual Analogue Scale".

SECONDARY OUTCOMES:
Mood of the patients | Measurements will be made before treatment, at the 1st week after treatment and at the 3rd month after treatment. Then change of the level of the mood of patients will be investigated.
  Mood of the patients will be determined by using "Beck Depression Scale".
Pressure pain threshold | Measurements will be made before treatment, at the 1st week after treatment and at the 3rd month after treatment. Then change of the level of pain pressure threshold will be investigated.
  Pressure pain threshold will be measured in patients using algometer.
Anxiety level of the patients | Measurements will be made before treatment, at the 1st week after treatment and at the 3rd month after treatment. Then change of the level of the anxiety will be investigated.
  Anxiety level of the patients will be determined by using "Beck Anxiety Scale"
Quality of life of the patients | Measurements will be made before treatment, at the 1st week after treatment and at the 3rd month after treatment. Then change of the quality of life will be investigated.
  Anxiety level of the patients will be determined by using "Short Form-36 Quality of Life. Scale"
Kinesiophobia of the patients | Measurements will be made before treatment, at the 1st week after treatment and at the 3rd month after treatment. Then change of the level of kinesiophobia will be investigated.
  Anxiety level of the patients will be determined by using "Tampa Kinesiophobia Scale".
Disability level of the patients | Measurements will be made before treatment, at the 1st week after treatment and at the 3rd month after treatment. Then change of the level of disablity will be investigated.
  Disability level of the patients will be determined by using "Neck Disability Questionnaire".
Global Assesment of the patients | The Global Assessment Scale will be used to evaluate patients at the 1st and 12th weeks after treatment.
  Global Assesment of the patients will be determined by using "Global Assessment Scale".

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep Karakuzu Güngör, MD, Principal Investigator — Ahi Evran Unıversity Faculty of Medicine; Fatmanur Aybala Koçak, MD, Study Director — Ahi Evran Unıversity Faculty of Medicine
Locations (1):
- Ahi Evran University Education and Research Hospital, Kırşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I believe that the study results will be beneficial to the world of science.

REFERENCES:
- [Background] Ong J, Claydon LS. The effect of dry needling for myofascial trigger points in the neck and shoulders: a systematic review and meta-analysis. J Bodyw Mov Ther. 2014 Jul;18(3):390-8. doi: 10.1016/j.jbmt.2013.11.009. Epub 2013 Nov 9. PMID 25042309